CLINICAL TRIAL: NCT03206034
Title: Stylistic Memory Enhancement
Acronym: SME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Nancy Chiaravalloti, Director Neuropsychology and Neuroscience Research, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E-769-13
Record Dates: First submitted 2017-06-27; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Multiple Sclerosis
Keywords: Memory; Cognition
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Double blind placebo controlled randomized control trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): The experimental group will meet with a study team member twice a week for 4 weeks (8 sessions) and receive memory strategy training.
  Interventions: Behavioral: Stylistic Memory Enhancement
- Control (Placebo Comparator): The control group participants will meet with a study team member twice a week for 4 weeks (8 sessions) and receive control memory exercises.
  Interventions: Behavioral: Stylistic Memory Enhancement

INTERVENTIONS:
Behavioral: Stylistic Memory Enhancement

SUMMARY:
Impairments in higher level cognitive processing, such as new learning and memory, are common in Multiple Sclerosis (MS) and negatively impact multiple aspects of everyday life, including occupational and social functioning. Despite this, few studies have attempted to remediate these cognitive deficits in order to improve everyday functioning. While not applied in traditional rehabilitation protocols as of yet, many techniques from cognitive psychology significantly improve learning and memory in healthy persons. These techniques include the generation effect (GE), the spacing effect (SE), and the testing effect (TE). These techniques have recently been incorporated into an 8-session treatment protocol, Stylistic Memory Enhancement (SME), designed to teach participants about each of the techniques, train them on how to apply the techniques in daily life and practice their application to daily life memory demanding situations. The protocol includes teaching participants how to restructure a memory demanding situation in order to make optimal use of self-generation, spaced learning and self-testing. The objective of the study is to test the efficacy of the SME in an MS population.

ELIGIBILITY:
Inclusion Criteria:

Clinically definite MS between the ages of 18 and 59. Participants must have impairment in new learning (determined by an in-person screen) with intact language comprehension.

Exclusion Criteria:

* History of alcohol or drug abuse/dependence,
* Major psychiatric disturbance (e.g. bipolar disorder, schizophrenia) and neurological history other than MS.
* Corticosteroid use within the last month prior to the participation.
* Less than 1 month post most recent exacerbation.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
California Verbal Learning Test (CVLT-II- Total learning | Baseline and post-intervention (5 weeks between testing sessions)
  Measure of change in new learning

SECONDARY OUTCOMES:
Memory Functioning Questionnaire | Baseline and post-intervention ( 5 weeks between testing sessions)
  Measure of change in Self-report of everyday memory functioning

IPD SHARING:
Plan to Share IPD: No